CLINICAL TRIAL: NCT03951103
Title: A Chart Review Study of Patients With Haemophilia A With Inhibitors Treated With rFVIIIFc (Elocta®) for Immune Tolerance Induction
Brief Title: rFVIIIFc (Elocta®) ITI Chart Review in Patients With Haemophilia A
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.Elocta-004
Record Dates: First submitted 2018-09-19; First posted 2019-05-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemophilia A With Inhibitor
Keywords: Elocta; rFVIIIFc
MeSH Terms: interventions — factor VIII-Fc fusion protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophili A patients: Patients treated with rFVIIIFc for ITI
  Interventions: Other: rFVIIIFc

INTERVENTIONS:
Other: rFVIIIFc — Drug according to prescription
  Other Names: Elocta

SUMMARY:
A chart review study of patients with haemophilia A with inhibitors treated with rFVIIIFc (Elocta®) for immune tolerance induction.

DETAILED DESCRIPTION:
A multicenter, international, non- interventional, retrospective and prospective medical chart review study. Data will be collected from medical records for patients diagnosed with haemophilia A who have been, or who are currently, treated with rFVIIIFc for ITI . The study will be descriptive in nature and report on baseline characteristics, treatment and outcomes for patients who have been, or who are currently, treated with rFVIIIFc for ITI.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with haemophilia A who have been, or who are currently, treated with rFVIIIFc for ITI.
* Signed and dated informed consent provided by the patient, or the patient's legally acceptable representative for patients under the legal age, before any study-related data collection are undertaken. Assent should be obtained from paediatric patients according to local regulations.

Exclusion Criteria:

* Current participation in any investigational medicinal product trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All haemophilia A patients who have been, or who are currently treated with rFVIIIFc for ITI meeting the inclusion and not meeting the exclusion criteria will be invited to participate. Approximately 45 patients from Europe and the Middle East are expected to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
ITI with rFVIIIFc: Main dose | From 2018 to 2022
  Main dose will be assessed on the prescribed dose (IU/kg)
ITI with rFVIIIFc: Main injection frequency | From 2018 to 2022
  Main injection frequency will be assessed on the prescribed frequency
ITI with rFVIIIFc: Duration | From 2018 to 2022
  Number of treatment months
ITI with rFVIIIFc: Concomitant by-passing agents | From 2018 to 2022
  Product name and main dose will be used to describe any concomitant use of by-passing agents.
Outcome of ITI with rFVIIIFc: Overall outcome | From 2018 to 2022
  The Investigator will assess overall outcome as: success, partial success, failure, early withdrawal or other.
Outcome of ITI with rFVIIIFc: Time to undetectable inhibitor titer | From 2018 to 2022
  Treatment time to reach undetectable inhibitor levels (<0.6 BU/ml)
Outcome of ITI with rFVIIIFc: Time to normal recovery | From 2018 to 2022
  Treatment time to reach normal recovery levels (≥66% of the expected value)
Outcome of ITI with rFVIIIFc: Time to success | From 2018 to 2022
  Treatment time to reach success (see outcome #5)
Outcome of ITI with rFVIIIFc: Inhibitor titer levels | From 2018 to 2022
  BU/ml
Outcome of ITI with rFVIIIFc: Half-life | From 2018 to 2022
  FVIII half-life (hours)
Outcome of ITI with rFVIIIFc: Recovery level | From 2018 to 2022
  FVIII recovery level (%)
Outcome of ITI with rFVIIIFc: Bleeds | From 2018 to 2022
  Number of bleeds per month during ITI-treatment
Long-term outcome after ITI with rFVIIIFc: Occurrence of relapse | From 2018 to 2022
  Occurrence of relapse (Yes/No) will be assessed by the investigator.
Long-term outcome after ITI with rFVIIIFc: Time to relapse | From 2018 to 2022
  Time to occurrence of relapse (see outcome #13)
Long-term outcome after ITI with rFVIIIFc: Treatment regimen | From 2018 to 2022
  Treatment regimen will be described as: ITI, prophylaxis or on-demand; and also by product used.
Long-term outcome after ITI with rFVIIIFc: Bleeds | From 2018 to 2022
  Number of bleeds per month.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lethagen, Study Director — Swedish Orphan Biovitrum
Locations (18):
- France (3):
  - Swedish Orphan Biovitrum Research Site, Paris
  - Swedish Orphan Biovitrum Research Site, Rennes
  - Swedish Orphan Biovitrum Research Site, Tours
- Germany (4):
  - Swedish Orphan Biovitrum Research Site, Frankfurt
  - Swedish Orphan Biovitrum Research Site, Friedrichshain
  - Swedish Orphan Biovitrum Research Site, Hanover
  - Swedish Orphan Biovitrum Research Site, Mitte
- Swedish Orphan Biovitrum Research Site, Dublin, Ireland
- Italy (4):
  - Swedish Orphan Biovitrum Research Site, Catania
  - Swedish Orphan Biovitrum Research Site, Catanzaro
  - Swedish Orphan Biovitrum Research Site, Genova
  - Swedish Orphan Biovitrum Research Site, Napoli
- Swedish Orphan Biovitrum Research Site, Kuwait City, Kuwait
- Swedish Orphan Biovitrum Research Site, Oslo, Norway
- Saudi Arabia (3):
  - Swedish Orphan Biovitrum Research Site, Riyadh
  - Swedish Orphan Biovitrum Research Site (a), Riyadh
  - Swedish Orphan Biovitrum Research Site (p), Riyadh
- Swedish Orphan Biovitrum Research Site, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klamroth R, Al Saleh M, Glosli H, Schiavulli M, Guillet B, Bystricka L, Schonstein A, Lethagen S. Immune Tolerance Induction With a Recombinant Factor VIII Fc in Haemophilia A: Data From a Chart Review Study. Eur J Haematol. 2025 Aug;115(2):134-141. doi: 10.1111/ejh.14427. Epub 2025 Apr 27. PMID 40289300